CLINICAL TRIAL: NCT06235268
Title: Prospective and Multicenter Italian Registry of Locally Advanced-Metastatic Urothelial Carcinoma (Saturno Study)
Brief Title: Prospective and Multicenter Italian Registry of Locally Advanced-Metastatic Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federation of Italian Cooperative Oncology Groups (Other)
Responsible Party: Sponsor
Other Study IDs: SATURNO
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Urothelial
MeSH Terms: conditions — Carcinoma | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Active systemic or non-systemic treatment (palliative or observation procedure) — The study includes medical visits and clinical-radiological re-evaluations according to clinical practice. The clinician will establish the number of visits necessary for each patient according to the needs encountered and depending on the treatment chosen.

SUMMARY:
Prospective and multicenter Italian registry intended for naïve adult patients affected by locally advanced-metastatic urothelial carcinoma intended for systemic treatment, or for palliative or observation procedures

DETAILED DESCRIPTION:
This is a multicentre, prospective and non-interventional study in which all patients treated according to clinical practice will be included. The registry will include all patients with metastatic urothelial carcinoma or with lymph node involvement defined as unsuitable for surgery. The study involves medical visits and clinical-radiological re-evaluations according to clinical practice. There are no additional procedures. The clinician will establish the number of visits necessary for each patient according to the needs encountered and depending on the treatment chosen. The participating centers were selected in such a way as to adequately represent all the different geographical areas. The duration of the study is 24 months: 12 months of enrollment plus 12 months of further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Cytological and/or histological diagnosis of urothelial carcinoma or at least with one urothelial component originating from the genitourinary tract.
* Radiological diagnosis of metastatic or locally advanced disease inoperable
* Primary bladder, ureter, renal pelvis and of the urethra are included
* No previous chemotherapy for advanced urothelial carcinoma or metastatic disease
* Age over 18 years old
* Ability to understand and sign the informed consent
* Patients for whom the clinician has opted for a therapeutic path not including active systemic treatments (iter palliative or observation) with certain diagnosis of metastatic disease
* Patients with lymph node extension of the disease who are not candidates to neoadjuvant treatment
* Any ECOG PS and therapeutic management is permitted.
* Previous surgeries and antineoplastic treatments are permitted as long as not carried out for metastatic disease (adjuvant and/or neoadjuvant)

Exclusion Criteria:

* Patients who have received previous systemic treatment for metastatic disease
* Patients with histological and/or cytological diagnosis without urothelial component
* Patients with muscle-infiltrating disease without evidence of metastatic disease
* Patients with non-muscle infiltrating disease without evidence of metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include all patients with metastatic urothelial carcinoma or with lymph node involvement defined as unsuitable for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Survival from Diagnosis to time of death
Progression free survival | up to 2 years
  the time from assignment to treatment to disease progression or death from any cause
Toxicities | up to 2 years
  Safety parameters commonly used for evaluating investigational systemic anticancer treatments are included as safety endpoints including, but not limited to, the incidence of, causality, and outcome of AEs/SAEs; and changes in vital signs and laboratory values. AEs will be assessed as defined by CTCAE, Version [5.0].
Treatment reality in Italy | over 2 years
  description of treatments selected for patients per line of therapy over the course of the project

CONTACTS AND LOCATIONS:
Locations (51):
- Italy (51):
  - Azienda Ospedaliera Universitaria delle Marche, Ancona
  - Ospedale Cardinal Massaia, Asti
  - Centro Regionale Oncologico di Aviano, Aviano
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Policlinico Universitario di Bari, Bari
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Spedali Civili, Brescia
  - Azienda Ospedaliera per l'Emergenza Cannizzaro, Catania
  - ASST Cremona, Cremona
  - Azienda Ospedaliera Universitaria Carreggi, Florence
  - Azienda Ospedaliero-Universitaria, Policlinico Riuniti, Foggia
  - Istituto Oncolgico Romagnolo di Meldola, Forlì
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Villa Scassi ASL 3 Genova, Genova
  - Casa della Salute, Aprilia, Latina
  - Ospedale Vito Fazzi, Lecce
  - ASST OVEST Milanese - Ospedale di Legnano, Legnano
  - IRCCS Fondazione istituto Nazionale dei Tumori, Milan
  - Humanitas Research Hospital Rozzano, Milan
  - Istituto Europeo di Oncologia (IEO), Milan
  - MultiMedica Sesto san Giovanni, Milan
  - Ospedale Civile Ramazzini di Carpi, Modena
  - Azienda Ospedaliera di Rilievo Nazionale Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - IRCCS Istituto Oncologico Veneto IOV, Padua
  - Ospedali di Cittadella e Camposampiero, ULSS 6 Euganea, Padua
  - Presidio Ospedaliero Andrea Tortora di Pagani, Pagani
  - Azienda di rilievo nazionale e di Alta Specializzazione (ARNAS) Civico, Palermo
  - Azienda Ospedaliero-Universitaria Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedali Riuniti Marche Nord, Pesaro
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Nuovo Ospedale di Prato "Santo Stefano", Azienda USL Toscana Centro, Prato
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - IRCCS Istituto Nazionale Tumori Regina Elena Roma, Roma
  - Ospedale Santa Maria Goretti, Roma
  - Policlinico Universitario Campus Bio-Medico, Roma
  - IRCCS Casa Sollievo della Sofferenza - San Giovanni Rotondo, San Giovanni Rotondo
  - Ospedale San Paolo Savona, Savona
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - A.O Ordine Mauriziano, Torino
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza, Torino
  - IRCCS Fondazione del Piemonte per l'Oncologia Candiolo, Torino
  - Ospedale S. Chiara, Trento
  - Azienda Sanitaria Universitaria Friuli Centrale - Ospedale "Santa Maria della Misericordia", Udine
  - Ospedale Michele e Pietro Ferrero, ASL CN2, Verduno
  - AULSS 8 Berica, Vicenza

IPD SHARING:
Plan to Share IPD: No